CLINICAL TRIAL: NCT02896608
Title: Neuronal Excitability of Hyperpolarization-activated Cyclic Nucleotide-gated (HCN1) Channel Mutations in Dravet Syndrome
Brief Title: Neuronal Excitability of HCN1 Channel Mutations in Dravet Syndrome
Acronym: EXCIDRAH
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: AGN_2015_11
Record Dates: First submitted 2016-08-23; First posted 2016-09-12 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Dravet Syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Dravet syndrome - HCN1 channel mutation: early infantile epileptic encephalopathy with HCN1 channel mutation
  Interventions: Device: measure of neuronal excitability
- control with epilepsy
  Interventions: Device: measure of neuronal excitability
- control without epilepsy
  Interventions: Device: measure of neuronal excitability

INTERVENTIONS:
Device: measure of neuronal excitability

SUMMARY:
This study addresses the changes in the axonal excitability parameters. It will compare these changes in patients with early infantile epileptic encephalopathy with HCN1 channel mutation and in control patients, with and without epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* early infantile epileptic encephalopathy with HCN1 channel mutation
* control patients with no neurologic pathology (age, gender and body temperature matched)
* epileptic patients (age, gender and body temperature matched)

Exclusion Criteria:

* pregnant or breast feeding patient

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with Dravet syndrome and control patients with and without epilepsy.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
hyperpolarizing electrotonus | baseline
hyperpolarizing threshold current | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France